CLINICAL TRIAL: NCT03330717
Title: Interventional Study on the Impact of the Hypnosis Used as Sedation or Relaxation (Virtual Reality) in the Breast Oncologic Surgery
Brief Title: Interventional Study on the Impact of the Hypnosis Used as Sedation or Relaxation in the Breast Oncologic Surgery
Acronym: OncoHypnose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/08JUL/311
Record Dates: First submitted 2017-10-19; First posted 2017-11-06 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General anesthesia (Placebo Comparator): Patients will undergo oncologic breast surgery on general anesthesia.
  Interventions: Procedure: General anesthesia
- Hypnosis sedation (Experimental): Patients will undergo oncologic breast surgery on hypnosis sedation.
  Interventions: Procedure: Hypnosis sedation
- General anesthesia with preoperative session of hypnosis (Experimental): Patients interested in hypnosis but too anxious to have surgery while on hypnosis sedation will undergo surgery on general anesthesia but will have a preoperative session of hypnosis relaxation using technology of virtual reality
  Interventions: Procedure: General anesthesia with preoperative session of hypnosis

INTERVENTIONS:
Procedure: General anesthesia — Patients will undergo oncologic breast surgery on general anesthesia.
  Arms: General anesthesia
Procedure: Hypnosis sedation — Patients will undergo oncologic breast surgery on hypnosis sedation.
  Arms: Hypnosis sedation
Procedure: General anesthesia with preoperative session of hypnosis — Patients will undergo surgery on general anesthesia but will have a preoperative session of hypnosis relaxation.
  Arms: General anesthesia with preoperative session of hypnosis

SUMMARY:
The aims of the study are to compare the recovering period between a group of patients with conventional sedation, a group using hypnosis as sedation during the surgery and a third group using hypnosis as a relaxation method and preparation but enjoying a classic sedation for their surgery.

Comparaison of pain ( different types of pain), consumption of pain killers ,anxiety and fatigue on day0,1, 8 after surgery and every. 3 months during the first 2 years of follow up.

Comparisons are also performed in substudies defined by treatments modalités. Inflammatory parameters s ( CRP_ C reactive protein, NLR- ( neutrophils to lymphocyte ratio) are measured on Day 0, 1, 8 and also salivary Immunoglobulins and different endocannabinoids.

DETAILED DESCRIPTION:
Hypnosis has already demonstrated benefits among breast cancer patients undergoing oncologic surgery. Different side effects were measured during the post operative period and at each follow up visit by physicians in order to carefully compare side effects in the 3 armes of patients..

Our hypothesis was that hypnosis sedation generates less perioperative inflammatory reaction.

A substudy of 50 patients was also dedicated to the investigation ofsalivary immunoglobulins and dosage of differents endocannabinoids

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Signed informed consent form
* Patient has to be in possession of her administrative laws and affiliated to the social security insurance.
* The patient must have a diagnosis of resectable breast cancer (in situ or invasive breast cancer). . Surgical procedure must include evaluation of the axillary area (sentinel lymph node biopsy and or axillary dissection)

Exclusion Criteria:

* Patient under 18 years old
* No signed informed consent form
* Patients who haven't her social security insurance and prisoners are not eligible.
* No evaluation of the axillary area.
* Breast cancer in men

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women with breast cancer will be included
Enrollment: 284 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of the days spent at the hospital post-surgery between the three groups | Day 0, 1, 8 and every 3 months for 2 years after surgery
  The aim of the study is to compare the recovering period hospitalisation and the different side effects (pain, anxiety, fatigue and consumption of pain killers ) during the post opérative period ( day 0, 1, 8- and at each follow up visit) between a group of patients with conventional sedation, a group using hypnosis as sedation during the surgery and a third group using hypnosis as a relaxation method and preparation but enjoying a classic sedation for their surgery
Comparaison of inflammatory parameters measured on day 0,1,8: CRP ( c reactive protein) and NLR ( neutrophils to lymphocyte ratio) | Day 0, 1, 8
  Blood test performed

SECONDARY OUTCOMES:
Substudy evaluation of salivary immunoglobulins and endocannabinoids among 50 patients (25 under general anesthesia and 25 under hypnosis sedation | Simples collected on Day 0, 1 and 8 for endocannabinoids and salivary simples collected on Day 0 and 8
  Blood and salivary simples to observe if hypnosis modifies salivary parameters and endocannabinoids system

CONTACTS AND LOCATIONS:
Overall Officials: Martine Berlière, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (2):
- Belgium (2):
  - Hôpital de Jolimont, Haine-Saint-Paul, Hainaut
  - Cliniques Universitaires Saint-Luc, Brussels